| A randomized control trials of web-based Educational program promoting response a | nd |
|---|---|
| willingness to handle elderly abuse among Gerontolgical nurses. | |

**IRB:** 91-c

Registration date: 16-1-2024

**Introduction:** 

Elderly abuse is a pervasive and concerning issue, particularly as the global population ages. Gerontological nurses play a pivotal role in identifying, preventing, and responding to elder abuse. However, there is a recognized need for targeted educational interventions to enhance nurses' knowledge, response efficacy, and willingness to address elder abuse effectively. This randomized controlled trial (RCT) aims to evaluate the impact of a web-based educational program designed to promote the response and willingness of gerontological nurses in handling elderly abuse cases. By employing a rigorous experimental design, this research seeks to contribute evidence-based insights that can inform educational strategies to empower nurses in safeguarding the well-being of elderly individuals.

# Methodology:

## 1. Study Design:

This research employs a randomized controlled trial design to assess the effectiveness of the webbased educational program. Participants will be randomly assigned to either the intervention group, receiving the educational program, or the control group with no intervention.

## 2. Participants:

The study will recruit a sample of gerontological nurses from diverse healthcare settings. Inclusion criteria include active employment as gerontological nurses, consent to participate, and access to the internet.

## 3. Intervention:

The web-based educational program will cover topics such as recognizing signs of elder abuse, understanding the psychological and physical impact on older adults, legal and ethical

considerations, and effective communication strategies. The intervention group will have access to the program for a specified period, while the control group will continue with standard practices.

### 4. Randomization:

Randomization will be conducted using computer-generated random numbers to ensure that participants are equally distributed between the intervention and control groups, minimizing selection bias.

#### 5. Outcome Measures:

The primary outcome measures include an assessment of participants' knowledge of elder abuse, response efficacy, and willingness to intervene. Pre- and post-intervention surveys, as well as follow-up assessments, will be conducted to evaluate the sustained impact of the educational program.

#### 6 Data Collection:

Data will be collected through self-administered surveys distributed electronically. The surveys will include validated instruments to measure knowledge levels, attitudes, and perceived efficacy related to handling elder abuse.

## 7. Statistical Analysis:

Descriptive statistics will be used to summarize participant characteristics. Between-group differences in knowledge, response efficacy, and willingness to handle elder abuse will be analyzed using appropriate statistical tests, such as t-tests or chi-square tests. Additionally, longitudinal analysis will be performed to assess the sustainability of the program's effects over time.

### 8. Ethical Considerations:

The study will adhere to ethical principles, obtaining informed consent from participants, ensuring confidentiality, and obtaining ethical approval from relevant institutional review boards.

By employing this robust methodology, the study aims to contribute valuable insights into the efficacy of web-based educational programs in enhancing gerontological nurses' preparedness and willingness to address elderly abuse, thereby promoting the overall well-being of the aging population.